CLINICAL TRIAL: NCT03911869
Title: A Phase 2, Open-Label, Randomized, Multicenter Trial of Encorafenib + Binimetinib Evaluating a Standard-dose and a High-dose Regimen in Patients With BRAFV600-Mutant Melanoma Brain Metastasis
Brief Title: An Open-Label, Randomized, Multicenter Trial of Encorafenib + Binimetinib Evaluating a Standard-dose and a High-dose Regimen in Patients With BRAFV600-mutant Melanoma Brain Metastasis
Acronym: POLARIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment of the target population. There were no safety, efficacy, or regulatory interaction involved in the decision to stop enrollment.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-818-201; C4221006 (Other: Alias Study Number); 2018-004555-21 (EudraCT Number)
Record Dates: First submitted 2019-03-14; First posted 2019-04-11 (Actual); Results first posted 2023-05-31 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Brain Metastases
Keywords: BRAFV600-mutant; melanoma; brain metastasis
MeSH Terms: conditions — Brain Neoplasms; Melanoma | interventions — encorafenib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Dose Arm (Experimental): Patients in the standard-dose treatment arm will receive encorafenib and binimetinib in 28-day cycles.
  * 450 mg encorafenib orally once a day (QD)
  * 45 mg binimetinib orally twice a day (BID)
  Patients who are able to tolerate the standard dose during the first 4 weeks of treatment (Cycle 1) should be dose-escalated to 600 mg encorafenib QD plus 45 mg binimetinib BID provided they meet protocol-defined criteria.
  Interventions: Drug: encorafenib; Drug: binimetinib
- High Dose Arm (Experimental): Patients in the high-dose treatment arm will receive encorafenib and binimetinib in 28-day cycles.
  * 300 mg encorafenib orally twice a day (BID)
  * 45 mg binimetinib orally twice a day (BID)
  Interventions: Drug: encorafenib; Drug: binimetinib

INTERVENTIONS:
Drug: encorafenib — taken orally
Drug: binimetinib — taken orally

SUMMARY:
This is a multicenter, randomized open-label Phase 2 study to assess the safety, efficacy and pharmacokinetic (PK) of 2 dosing regimens of encorafenib + binimetinib combination in patients with BRAFV600-mutant melanoma with brain metastasis. Approximately 100 patients will be enrolled, including 9 patients in a Safety Lead-in of the high-dose treatment arm. After a Screening Period, treatment will be administered in 28-day cycles and will continue until disease progression, unacceptable toxicity, withdrawal of consent, start of subsequent anticancer therapy, death.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed diagnosis of cutaneous melanoma with metastases to the brain.
* Presence of B-RAF proto-oncogene, V600 mutant (BRAFV600) mutation in tumor tissue previously determined by a local PCR or NGS-based assay at any time prior to Screening or by a central laboratory during Screening.
* Must have at least 1 parenchymal brain lesion ≥ 0.5 cm and ≤ 4 cm, defined as a magnetic resonance imaging (MRI) contrast-enhancing lesion that may be accurately measured in at least 1 dimension. (Measurable intracranial lesions that have been previously irradiated and have not been shown to be progressing following irradiation should not be considered as target lesions).
* Patients may have received the following prior therapies:

  1. Safety Lead-in, Phase 2 Randomized , Phase 2 Arm A Cohort 1: May have received prior local therapy for brain metastases including but not restricted to brain surgery, whole brain radiotherapy, stereotactic radiotherapy or stereotactic radiosurgery. Multiple local (brain) therapies or combinations of local therapies are allowed. For patients receiving local therapy to all brain lesions (including WBRT), progression of pre-existing lesions based on RECIST 1.1 (> 20% increase in longest diameter on baseline scan) or new measurable lesions are required. For patients receiving local therapy for some but not all lesions, disease progression based on RECIST 1.1 is not required as long as there are remaining brain lesions that are measurable and not previously treated.
  2. Phase 2 Arm A Cohort 2: Received no prior local therapy (e.g., brain surgery, craniotomy, SRS or SRT) for brain metastases.
  3. All patients (Safety Lead-In and Phase 2): May have received prior immunotherapy.
  4. All patients (Safety Lead-In and Phase 2): If receiving concomitant corticosteroids must be on a stable or decreasing dose for at least 2 weeks prior to first dose of study treatment (up to a total daily dose of 4mg of dexamethasone or equivalent).
* An Eastern Cooperation Oncology Group Performance Status (ECOG PS) of 0 or 1 and Karnofsky score ≥ 80
* Adequate bone marrow, organ function and laboratory parameters

Key Exclusion Criteria:

* Patients with symptomatic brain metastasis.
* Uveal or mucosal melanoma.
* History of or current leptomeningeal metastases.
* Treatment with SRS or craniotomy within 14 days prior to start of study treatment, or treatment with whole-brain radiation within 28 days prior to study treatment. Patients who received local therapy should have complete recovery with no neurological sequelae.
* Either of the following:

  1. Radiation therapy to non-brain visceral metastasis within 2 weeks prior to start of study treatment;
  2. Continuous or intermittent small-molecule therapeutics or investigational agents within 5 half-lives of the agent (or within 4 weeks prior to start of study treatment, when half-life is unknown).
* Patients treated in the adjuvant setting with BRAF or MEK inhibitor(s) < 6 months prior to enrollment. Patients who received BRAF or MEK inhibitors in the metastatic setting are excluded.
* Patient has not recovered to ≤ Grade 1 from toxic effects of prior therapy before starting study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (11):
  - The Angeles Clinic And Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - The Retina Partners, Santa Monica, California
  - Rocky Mountain Lions Eye Institute (RMLEI), Aurora, Colorado
  - University of Colorado Denver CTO/CTRC - Outpatient., Aurora, Colorado
  - University of Colorado Hospital - Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion, Aurora, Colorado
  - University of Colorado Hospital, Aurora, Colorado
  - Oregon Health & Science University Center for Health & Healing 2, Portland, Oregon
  - OHSU Center for Health and Healing, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Argentina (3):
  - Instituto Médico Especializado Alexander Fleming, Buenos Aires, Ciudad Autónoma de Buenosaires
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Fundacion CIDEA, CABA
- Australia (4):
  - Crows Nest Eye Surgery, Crows Nest, New South Wales
  - Melanoma Institute Australia, North Sydney, New South Wales
  - Royal north shore center hospital dermatology clinics, St Leonards, New South Wales
  - Mater Imaging, Wollstonecraft, New South Wales
- UZ Antwerpen, Edegem, Antwerpen, Belgium
- Italy (6):
  - Azienda Universitaria Policlinico Federico II, Napoli, Naples
  - S.C. Cardiologia, Napoli
  - S.C. Farmacia, Napoli
  - S.C. Medicina Nucleare e Terapia Metabolica, Napoli
  - SC Melanoma, Immunoterapia Oncologica e Terapie Innovative, Napoli
  - U.O. Radiodiagnostica 1, Napoli

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-818-201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study had 2 parts, Safety lead-in and Phase 2. In Phase 2, participants would be randomized either to the standard-dose or high-dose treatment, only if high dose was determined to be safe in safety lead-in.
Pre-assignment Details: Pfizer and the Steering Committee reviewed safety lead-in data and decided not to evaluate high dose combination of encorafenib + binimetinib in Phase 2 of the study.
Groups:
- Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID: Participants diagnosed with BRAFV600-mutant melanoma brain metastasis received combination therapy of encorafenib (300 milligram [mg] orally, twice daily [BID]) and binimetinib (45 mg orally, BID) in 28-day cycles and continued until disease progression, unacceptable toxicity, withdrawal of consent, start of subsequent anticancer therapy, or death, whichever occurred first. Participants were followed up to 30 days after last dose of study drug.
- Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID: Participants diagnosed with BRAFV600-mutant melanoma brain metastasis received standard combination therapy of encorafenib (450 mg orally, once daily [QD]) and binimetinib (45 mg orally, BID) in 28-day cycles and participants who were able to tolerate the encorafenib 450 mg dose further received 600 mg QD after 4 Weeks. Participants were followed up to 30 days after last dose of study drug.
- Phase 2, High Dose Arm: Encorafenib 300 mg BID + Binimetinib 45 mg BID: If high dose in safety lead-in was determined safe then participants were to be randomized in high dose arm in Phase 2 to receive combination therapy of encorafenib (300 mg orally, BID), and binimetinib (45 mg orally, BID) in 28-day cycles until disease progression, unacceptable toxicity, withdrawal of consent, start of subsequent anticancer therapy, or death, whichever occurred first.
Period: Safety Lead-in Phase
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID | Phase 2, High Dose Arm: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Started | 10 | 0 | 0 (High dose was not determined safe, hence no participants randomized into this arm.)
Completed | 0 | 0 | 0
Not Completed | 10 | 0 | 0
Not completed — Death | 7 | 0 | 0
Not completed — Study termination by sponsor | 2 | 0 | 0
Not completed — Other | 1 | 0 | 0
Period: Phase 2
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID | Phase 2, High Dose Arm: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Started | 0 | 3 (Participants entered in Phase 2 were included in this period.) | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 3 | 0
Not completed — Death | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received at least 1 dose of any study drug.
Groups:
- Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID: Participants diagnosed with BRAFV600-mutant melanoma brain metastasis received combination therapy of encorafenib (300 mg orally, BID) and binimetinib (45 mg orally, BID) in 28-day cycles and continued until disease progression, unacceptable toxicity, withdrawal of consent, start of subsequent anticancer therapy, or death, whichever occurred first. Participants were followed up to 30 days after last dose of study drug.
- Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID: Participants diagnosed with BRAFV600-mutant melanoma brain metastasis received standard combination therapy of encorafenib (450 mg orally, QD) and binimetinib (45 mg orally, BID) in 28-day cycles and participants who were able to tolerate the encorafenib 450 mg dose further received 600 mg QD after 4 Weeks. Participants were followed up to 30 days after last dose of study drug.
- Total: Total of all reporting groups
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID | Total
Number analyzed (Participants) | 10 | 3 | 13
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.2 (12.94) | 45.7 (5.86) | 59.2 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 8 | 2 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 3 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs): Safety Lead-in (SLI) Phase
Description: DLT: any adverse event (AE) or laboratory abnormality not explained by underlying disease/disease progression/intercurrent illness/concomitant therapies/resulting in inability to tolerate 75% of planned dose of binimetinib or encorafenib during Cycle 1. Left ventricular ejection fraction (LVEF) >10%, Grade (G)>=3 cardiac disorders; G3/4 hypertension vascular disorders; G3/4 rash, hand foot skin reaction, photosensitivity; G3/4 diarrhea, nausea/vomiting Total bilirubin (TBL) G>=3 (>3.0*upper limit of normal [ULN)]);AST/ALT>5-8*ULN>5 days,>8*ULN,>3*ULN concurrent TBL>2*ULN;G>=3 serum creatinine, CK elevation, ECG QTcF prolonged,G3 troponin, electrolyte>72 hours,G3/4 amylase/lipase.G4 ANC, platelet count>7 days;G3/4 platelet count, other AE except lymphopenia. G>=3 retinopathy, other disorder>21 days; G2 uveitis/eye pain/blurred vision/decreased visual acuity; G4 other disorder; Other hematologic/non hematologic G>=3 AE. This outcome measure was planned to be analyzed in SLI phase only.
Time Frame: Cycle 1 of SLI phase (up to 28 days)
Population: The dose-determining set included all participants enrolled in the high-dose treatment arm in the safety lead-in who completed one 28-day cycle of treatment and received at least 75 percentage (%) of the planned cumulative dose of both study drugs or discontinued treatment because of DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 9
Participants | 3

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events Graded by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI _CTCAE) Version (v) 4.03: SLI Phase
Description: AE: any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs: events between first dose of study drug up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state or start of subsequent anticancer drug therapy minus 1 day, whichever occurred first. Grades by NCI CTCAE v.4.03: Grade 1= asymptomatic or mild , clinical or diagnostic observations only, intervention not indicated; Grade 2= moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3= severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4= life-threatening consequence, urgent intervention indicated; Grade 5= death related to AE. Number of participants with AEs per maximum grades were reported.
Time Frame: Day 1 of dosing up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: The safety set included all participants who received at least 1 dose of any study drug. This outcome measure was planned to be analyzed in SLI phase only.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  Grade 1 | 1
  Grade 2 | 3
  Grade 3 | 5
  Grade 4 | 1
  Grade 5 | 0

3. Primary Outcome: Number of Participants With Hepatology Laboratory Test Abnormalities: SLI Phase
Description: Hepatology laboratory abnormalities included following parameters: alanine aminotransferase (ALT), aspartate aminotransferase (AST), ALT or AST greater than or equal to (>=) 3*upper limit normal (ULN), >=5*ULN, >=10*ULN, >=20*ULN; total bilirubin (TBILI): >=2*ULN; ALT >=3*ULN and TBILI >=2*ULN; AST >=3*ULN and TBILI >=2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN and ALP >2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN and ALP <=2*ULN or missing. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  ALT: >=3*ULN | 3
  ALT: >=5*ULN | 1
  AST: >=3*ULN | 3
  ALT or AST: >=3*ULN | 3
  ALT or AST: >=5*ULN | 1

4. Primary Outcome: Number of Participants With Shift From Baseline for Hematology and Coagulation Laboratory Test Abnormalities Based on NCI-CTCAE v4.03: SLI Phase
Description: Hematology and coagulation laboratory test included: activated partial thromboplastin time prolonged, anemia, hemoglobin increased, international normalized ratio (INR) increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, and white blood cell decreased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Grade 0 was assigned for all non-missing values not graded as 1 or higher per CTCAE criteria. Number of participants with shift from baseline for hematology and coagulation laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: The safety set included all participants who received at least 1 dose of any study drug. Here, "Number Analyzed" signifies participants evaluable for specified rows. This outcome measure was planned to be analyzed in SLI phase only.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 6
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 0 (post-baseline) | 5
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 6
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Anemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Anemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 7
  Anemia: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Hemoglobin increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  INR increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Leukocytosis: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 2 (post-baseline) | 2
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 3 (post-baseline) | 3
  Lymphocyte count increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 8
  Lymphocyte count increased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 9
  Lymphocyte count increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Neutrophil count decreased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 9
  Neutrophil count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 8
  Neutrophil count decreased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 9
  Neutrophil count decreased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Platelet count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 7
  Platelet count decreased: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  White blood cell decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 8
  White blood cell decreased: Grade 0 (baseline) to Grade 2 (post-baseline) | 2

5. Primary Outcome: Number of Participants With Shift From Baseline for Biochemistry Laboratory Test Abnormalities Based on NCI-CTCAE v4.03: SLI Phase
Description: Biochemistry laboratory test included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, creatine kinase (CK) increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase increased, and serum amylase increased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Grade 0 was assigned for all non-missing values not graded as 1 or higher per CTCAE criteria. Number of participants with shift from baseline for biochemistry laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 8
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 8
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 8
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 2
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 8
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 3 (post-baseline) | 1
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 1 (post-baseline) | 2
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 8
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 5
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 8
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  Alkaline phosphatase increased: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Alkaline phosphatase increased: Grade 1 (baseline) to Grade 0 (post-baseline) | 2
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 8
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 4
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 8
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 8
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 2
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline) | 1
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 1 (post-baseline) | 1
  Blood bilirubin increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  CK increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 6
  CK increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  CK increased: Grade 0 (baseline) to Grade 4 (post-baseline) | 1
  Creatinine increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 9
  Creatinine increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Hypercalcemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hyperglycemia: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 8
  Hyperglycemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 5
  Hyperglycemia: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 8
  Hyperglycemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Hyperglycemia: Grade 0 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 8
  Hyperglycemia: Grade 0 (baseline) to Grade 3 (post-baseline) | 2
  Hyperglycemia: Baseline to post-baseline: number analyzed (Participants) | 2
  Hyperglycemia: Baseline to post-baseline | 1
  Hyperglycemia: Missing (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Hyperglycemia: Missing (baseline) to Grade 1 (post-baseline) | 1
  Hyperkalemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hypermagnesemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 9
  Hypermagnesemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Hypernatremia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hypoalbuminemia: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 9
  Hypoalbuminemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 6
  Hypoalbuminemia: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 9
  Hypoalbuminemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  Hypoalbuminemia: Grade 2 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 1
  Hypoalbuminemia: Grade 2 (baseline) to Grade 2 (post-baseline) | 1
  Hypocalcemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 8
  Hypocalcemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  Hypoglycemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hypokalemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hypomagnesemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 10
  Hyponatremia: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 8
  Hyponatremia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hyponatremia: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 8
  Hyponatremia: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  Hyponatremia: Grade 0 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 8
  Hyponatremia: Grade 0 (baseline) to Grade 3 (post-baseline) | 3
  Hyponatremia: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Hyponatremia: Grade 1 (baseline) to Grade 0 (post-baseline) | 1
  Hyponatremia: Grade 1 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 2
  Hyponatremia: Grade 1 (baseline) to Grade 3 (post-baseline) | 1
  Hypophosphatemia: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 7
  Hypophosphatemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 6
  Hypophosphatemia: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 7
  Hypophosphatemia: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Hypophosphatemia: Missing (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Hypophosphatemia: Missing (baseline) to Grade 0 (post-baseline) | 1
  Hypophosphatemia: Missing (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 2
  Hypophosphatemia: Missing (baseline) to Grade 2 (post-baseline) | 1
  Lipase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 7
  Lipase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 3
  Serum amylase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 10

6. Primary Outcome: Number of Participants With Notable Abnormal Vital Signs: SLI Phase
Description: Vital signs included: systolic and diastolic blood pressure (BP),pulse rate,weight and temperature.Systolic and diastolic BP was measured in millimeters of mercury (mmHg) based on criteria:High Systolic BP:>=160 mmHg and increase >=20 mmHg from baseline;High Diastolic BP:>=100 mmHg and increase>=15 mmHg from baseline;Low Systolic BP:<=90 mmHg with decrease from baseline of >=20 mmHg;Low Diastolic BP:<=50 mmHg with decrease from baseline of >=15 mmHg;Pulse rate was measured in beats per minute (bpm) based on criteria:High pulse rate >=120 bpm with increase from baseline of >=15 bpm;Low pulse rate <=50 bpm with decrease from baseline of >=15 bpm;Weight was measured in in kilogram (kg) based on criteria:Increase from baseline of >=10%,:>=20% decrease from baseline;Temperature was measured in degree Celsius (C) based on criteria:High body temperature >=37.5 degree C,Low body temperature <=36 degree C.Only those vital signs parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  High systolic BP | 2
  Low diastolic BP | 1
  High pulse rate | 1
  Low pulse rate | 1
  Increased body weight | 2
  High body temperature | 1
  Low body temperature | 3

7. Primary Outcome: Number of Participants With Notable Abnormal Electrocardiogram (ECG) Values: SLI Phase
Description: In this outcome measure, number of participants with notable abnormal ECG values included: Fridericia's Correction Formula (QTcF) values in millisecond (msec) based on following criteria: 1) Increase from baseline >30 msec; 2) Increase from baseline >60 msec; 3) New >450 msec; 4) New >480 msec; and 5) New >500 msec; heart rate values in bpm based on following criteria: 1) Increase from baseline >25% and to a value >100; 2) Decrease from baseline >25% and to a value <50. Only those ECG parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  QTcF: New >450 msec | 6
  QTcF:Increase from baseline >30 msec | 5
  QTcF:Increase from baseline >25% and to a value >100 | 1

8. Primary Outcome: Number of Participants With Incidence of Dose Interruptions, Dose Modifications and Discontinuations Due to AEs: SLI Phase
Description: An AE is any untoward medical occurrence in clinical investigation participant administered a product or medical device; event need not necessarily to have a causal relationship with treatment or usage. In this outcome measure, number of participants with incidence of dose interruptions, dose modifications and discontinuations due to AEs were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in SLI Phase, maximum duration up to 10.4 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Participants
  Dose interruptions due to AE | 6
  Dose modifications due to AE | 4
  Discontinuations due to AE | 1

9. Primary Outcome: Brain Metastasis Response Rate (BMRR) Based on Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (mRECIST v1.1): Phase 2
Description: BMRR was reported in terms of percentage of participants who achieved a confirmed best overall response (BOR) of confirmed complete response (CR) or partial response (PR) in brain metastasis per mRECIST v1.1 from date of first dose until disease progression, death due to any cause, or start of subsequent anticancer therapy, whichever occurred first. BOR: best response recorded from date of first dose of study treatment until progression by investigator assessment at each time point. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until disease progression, death due to any cause or subsequent therapy initiation, whichever occurred first in Phase 2 (approximately up to 8.3 months)
Population: The safety set included all participants who received at least 1 dose of any study drug. This outcome measure was planned to be analyzed in phase 2 only.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Percentage of participants | 66.7 [9.4 to 99.2]

10. Secondary Outcome: Extracranial Response Rate Based on RECIST v1.1: SLI Phase and Phase 2
Description: Extracranial response rate was defined as the percentage of participants with a BOR of confirmed CR or confirmed PR in extracranial lesions by investigator assessment per RECIST v1.1. BOR: best response recorded from date of first dose of study treatment until progression by investigator assessment at each time point. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of first dose until disease progression, death due to any cause or subsequent therapy initiation, whichever occurred first in SLI Phase (approximately up to 10.4 months) and Phase 2 (approximately up to 8.3 months)
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Percentage of participants | 60.0 [26.2 to 87.8] | 100 [29.2 to 100]

11. Secondary Outcome: Global Response Rate: SLI Phase and Phase 2
Description: Global response rate was defined as the percentage of participants with a BOR of confirmed CR or confirmed PR by investigator assessment in brain metastasis and extracranial lesions per combined mRECIST v1.1 and RECIST v1.1, respectively. BOR: best response recorded from date of first dose of study treatment until progression by investigator assessment at each time point. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum of the diameters (e.g., percent change from baseline).
Time Frame: as for outcome 10
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Percentage of participants | 50.0 [18.7 to 81.3] | 100 [29.2 to 100]

12. Secondary Outcome: Disease Control Rate (DCR) for Brain Metastasis Response Based on mRECIST v1.1: SLI Phase and Phase 2
Description: DCR was defined as the percentage of participants with a BOR of CR, PR or stable disease (SD) by Investigator assessment per mRECIST v1.1. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD). PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded since the treatment started.
Time Frame: as for outcome 10
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Percentage of participants | 100 [69.2 to 100] | 100 [29.2 to 100]

13. Secondary Outcome: DCR for Extracranial Response Based on RECIST v1.1: SLI Phase and Phase 2
Description: DCR was defined as the percentage of participants with a BOR of CR, PR or SD by Investigator assessment per RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum demonstrates an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered progression.
Time Frame: as for outcome 10
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Percentage of participants | 70.0 [34.8 to 93.3] | 100 [29.2 to 100]

14. Secondary Outcome: DCR for Global Response: SLI Phase and Phase 2
Description: DCR was defined as the percentage of participants with a BOR of CR, PR or SD by Investigator assessment per RECIST v1.1. CR: disappearance of all target lesions. Any pathological lymph nodes must be <10 mm on the short axis. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum of the diameters (e.g., percent change from baseline). SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to quality for PD. PD: at least a 20% increase in the sum of the diameters of target lesions, taking as a reference the smallest sum of diameters recorded since the treatment started (i.e., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of at least 5 mm.
Time Frame: as for outcome 10
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Percentage of participants | 90.0 [55.5 to 99.7] | 100 [29.2 to 100]

15. Secondary Outcome: Duration of Response (DOR) for Brain Metastasis Response Based on mRECIST v1.1: SLI Phase and Phase 2
Description: DOR: time from date of first radiographic response (CR or PR) to earliest documented disease progression or death due to any cause. CR: disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. DOR (months) = (date of event or censoring - date of first CR or PR + 1)/30.4375. If a participant with a CR or PR did not have an event at time of analysis cutoff or with an event more than 16 weeks (for first 11 cycles after treatment start date) or 24 weeks (after Cycle 11) after last adequate tumor assessment, participant was censored on date of last adequate tumor assessment that documented no progression.
Time Frame: From date of first radiographic response (CR or PR) to earliest documented disease progression or death due to any cause in SLI Phase (approximately up to 10.4 months) and Phase 2 (approximately up to 8.3 months)
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Months | 3.3 [2.8 to 8.5] | 5.6 [5.0 to 6.2]

16. Secondary Outcome: DOR for Global Response: SLI Phase and Phase 2
Description: DOR: time from date of first radiographic response (CR or PR) to earliest documented disease progression or death due to any cause. CR: disappearance of all target lesions. Any pathological lymph nodes must be <10 mm on the short axis. PR: at least a 30% decrease in the sum of the diameters of target lesions, taking as a reference the baseline sum of the diameters (e.g., percent change from baseline). DOR (months) = (date of event or censoring - date of first CR or PR + 1)/30.4375. If a participant with a CR or PR did not have an event at time of analysis cutoff or with an event more than 16 weeks (for first 11 cycles after treatment start date) or 24 weeks (after Cycle 11) after last adequate tumor assessment, participant was censored on date of last adequate tumor assessment that documented no progression.
Time Frame: as for outcome 15
Population: The safety set included all participants who received at least 1 dose of any study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Months | 2.9 [2.8 to 8.5] | 5.0 [3.9 to 6.2]

17. Secondary Outcome: DOR for Extracranial Response Based on RECIST v1.1: SLI Phase and Phase 2
Description: DOR: time from date of first radiographic response (CR or PR) to earliest documented disease progression or death due to any cause. CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. DOR (months) = (date of event or censoring - date of first CR or PR + 1)/30.4375. If a participant with a CR or PR did not have an event at time of analysis cutoff or with an event more than 16 weeks (for first 11 cycles after treatment start date) or 24 weeks (after Cycle 11) after last adequate tumor assessment, participant was censored on date of last adequate tumor assessment that documented no progression.
Time Frame: as for outcome 15
Population: The safety set included all participants who received at least 1 dose of any study drug. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for specified rows. Data has been presented per participant as data was not summarized due to due to limited number of participants with events.
Measure: Number; unit: Months
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 6 | 3
Months
  Participant 1: number analyzed (Participants) | 1 | 0
  Participant 1 | 2.4 |
  Participant 2: number analyzed (Participants) | 1 | 0
  Participant 2 | 4.3 |
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | 5.5 |
  Participant 4: number analyzed (Participants) | 1 | 0
  Participant 4 | 2.8 |
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 1.8 |
  Participant 6: number analyzed (Participants) | 1 | 0
  Participant 6 | 2.8 |
  Participant 7: number analyzed (Participants) | 0 | 1
  Participant 7 |  | 7.7
  Participant 8: number analyzed (Participants) | 0 | 1
  Participant 8 |  | 3.9
  Participant 9: number analyzed (Participants) | 0 | 1
  Participant 9 |  | 7.3

18. Secondary Outcome: Progression Free Survival (PFS) for Brain Metastasis Based on mRECIST v1.1: SLI Phase and Phase 2
Description: PFS was defined as the time from date of the first dose of study treatment to the earliest documented disease progression (PD) by Investigator assessment, or death due to any cause, whichever occurs first. PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters recorded since the treatment started (e.g., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase of at least 5 mm. If a participant did not had a PFS event at the time of the analysis cutoff or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment.
Time Frame: From date of first dose of study treatment to the earliest documented disease progression by investigator assessment, or death due to any cause, whichever occurs first in SLI (approximately up to 10.4 months) and Phase 2 (approximately up to 8.3 months)
Population: The safety set included all participants who received at least 1 dose of any study drug. Here, 'Number Analyzed' signifies participants evaluable for specified rows. Data has been presented per participant as data was not summarized due to due to limited number of participants with events.
Measure: Number; unit: Months
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Months
  Participant 1: number analyzed (Participants) | 1 | 0
  Participant 1 | 3.5 |
  Participant 2: number analyzed (Participants) | 1 | 0
  Participant 2 | 3.7 |
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | 3.6 |
  Participant 4: number analyzed (Participants) | 1 | 0
  Participant 4 | 5.5 |
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 9.4 |
  Participant 6: number analyzed (Participants) | 1 | 0
  Participant 6 | 3.7 |
  Participant 7: number analyzed (Participants) | 1 | 0
  Participant 7 | 3.8 |
  Participant 8: number analyzed (Participants) | 1 | 0
  Participant 8 | 7.3 |
  Participant 9: number analyzed (Participants) | 1 | 0
  Participant 9 | 3.7 |
  Participant 10: number analyzed (Participants) | 1 | 0
  Participant 10 | 5.4 |
  Participant 11: number analyzed (Participants) | 0 | 1
  Participant 11 |  | 7.4
  Participant 12: number analyzed (Participants) | 0 | 1
  Participant 12 |  | 5.5
  Participant 13: number analyzed (Participants) | 0 | 1
  Participant 13 |  | 6.8

19. Secondary Outcome: PFS for Global Tumor Assessment: SLI Phase and Phase 2
Description: PFS was defined as the time from date of the first dose of study treatment to the earliest documented disease progression (PD) by Investigator assessment, or death due to any cause, whichever occurs first. PD: at least a 20% increase in the sum of the diameters of target lesions, taking as a reference the smallest sum of diameters recorded since the treatment started (i.e., percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of at least 5 mm. Global tumor assessment consists of brain metastasis and extracranial lesions. If a participant did not had a PFS event at the time of the analysis cutoff or at the start of any new anticancer therapy, PFS was censored at the date of last adequate tumor assessment.
Time Frame: as for outcome 18
Population: The safety set included all participants who received at least 1 dose of any study drug. Here, 'Number Analyzed' signifies participants evaluable for specified rows. Data has been presented per participant as data was not summarized due to limited number of participants with events.
Measure: Number; unit: Months
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 10 | 3
Months
  Participant 1: number analyzed (Participants) | 1 | 0
  Participant 1 | 3.5 |
  Participant 2: number analyzed (Participants) | 1 | 0
  Participant 2 | NA — Participant has been censored at baseline for no adequate baseline assessment. |
  Participant 3: number analyzed (Participants) | 1 | 0
  Participant 3 | 3.6 |
  Participant 4: number analyzed (Participants) | 1 | 0
  Participant 4 | NA — Participant has been censored at baseline for no adequate baseline assessment. |
  Participant 5: number analyzed (Participants) | 1 | 0
  Participant 5 | 9.4 |
  Participant 6: number analyzed (Participants) | 1 | 0
  Participant 6 | 3.7 |
  Participant 7: number analyzed (Participants) | 1 | 0
  Participant 7 | 3.8 |
  Participant 8: number analyzed (Participants) | 1 | 0
  Participant 8 | 7.3 |
  Participant 9: number analyzed (Participants) | 1 | 0
  Participant 9 | 3.7 |
  Participant 10: number analyzed (Participants) | 1 | 0
  Participant 10 | 1.0 |
  Participant 11: number analyzed (Participants) | 0 | 1
  Participant 11 |  | 7.4
  Participant 12: number analyzed (Participants) | 0 | 1
  Participant 12 |  | 5.5
  Participant 13: number analyzed (Participants) | 0 | 1
  Participant 13 |  | 6.8

20. Secondary Outcome: BMRR Based on mRECIST v1.1: SLI Phase
Description: BMRR: percentage of participants who achieved a confirmed best overall response (BOR) of confirmed CR or PR in brain metastasis per mRECIST v1.1 from date of first dose until disease progression, death due to any cause, or start of subsequent anticancer therapy, whichever occurs first. BOR: best response recorded from date of first dose of study treatment until progression by investigator assessment at each time point. CR: Disappearance of all target lesions. PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters (e.g., percent change from baseline).
Time Frame: From date of first dose until disease progression, death due to any cause or subsequent therapy initiation, whichever occurred first in SLI Phase (approximately up to 10.4 months)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 10
Percentage of participants | 60.0 [26.2 to 87.8]

21. Secondary Outcome: Overall Survival: SLI Phase and Phase 2
Description: Overall survival (OS) was defined as the time from date of the first dose of study treatment to the date of death due to any cause. If a death was not observed by the date of the analysis cutoff, OS was censored at the date of last contact. OS (months) = (date of death or censoring - date of first dose +1)/30.4375
Time Frame: as for outcome 18
Population: Data was not collected due to the premature termination of the study and consequent lack of meaningful data, data are not available and no analyses were performed.
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Number of Participants With Treatment Emergent AEs of Maximum Severity Grades Based on NCI CTCAE v4.03: Phase 2
Description: AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship.TEAEs were events between 1st dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state or start of subsequent anticancer drug therapy minus 1 day, whichever occurs first.Severity was graded by NCI CTCAE v.4.03.Grade 1:asymptomatic or mild symptoms, clinical or diagnostic observations only, intervention not indicated;Grade 2:moderate, minimal, local or noninvasive intervention indicated, limiting age-appropriate instrumental ADL;Grade 3:severe or medically significant but not immediately life-threatening, hospitalization or prolongation of existing hospitalization indicated, disabling, limiting self-care ADL;Grade 4:life-threatening consequence, urgent intervention indicated; Grade 5:death related to AE. Only those categories in which at least 1 participant had data were reported.
Time Frame: Day 1 of dosing up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants
  Grade 2 | 2
  Grade 4 | 1

23. Secondary Outcome: Number of Participants With Hepatology Laboratory Test Abnormalities: Phase 2
Description: Hepatology laboratory abnormalities included following parameters: ALT, AST, ALT or AST >=3*ULN, >=5*ULN, >=10*ULN, >=20*ULN; TBILI: >=2*ULN; ALT >=3*ULN and TBILI >=2*ULN; AST >=3*ULN and TBILI >=2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN and ALP >2*ULN; ALT or AST >=3*ULN and TBILI >=2*ULN and ALP <=2*ULN or missing. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants
  ALT: >=3*ULN | 2
  ALT: >=5*ULN | 1
  ALT: >=10*ULN | 1
  ALT: >=20*ULN | 1
  AST: >=3*ULN | 1
  AST: >=5*ULN | 1
  AST: >=10*ULN | 1
  ALT or AST: >=3*ULN | 2
  ALT or AST: >=5*ULN | 1
  ALT or AST: >=10*ULN | 1
  ALT or AST: >=20*ULN | 1

24. Secondary Outcome: Number of Participants With Shift From Baseline for Hematology and Coagulation Laboratory Test Abnormalities Based on NCI-CTCAE v4.03: Phase 2
Description: Hematology and coagulation laboratory test included: activated partial thromboplastin time prolonged, anemia, hemoglobin increased, INR increased, leukocytosis, lymphocyte count decreased, lymphocyte count increased, neutrophil count decreased, platelet count decreased, and white blood cell decreased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Grade 0 was assigned for all non-missing values not graded as 1 or higher per CTCAE criteria. Number of participants with shift from baseline for hematology and coagulation laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: The safety set included all participants who received at least 1 dose of any study drug. Here, "Number Analyzed" signifies participants evaluable for specified rows. This outcome measure was planned to be analyzed in phase 2 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 1
  Activated partial thromboplastin time prolonged: Grade 0 (baseline) to Grade 0 (post-baseline) | 1
  Anemia: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Anemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Anemia: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 2
  Anemia: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Anemia: Grade 1 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 1
  Anemia: Grade 1 (baseline) to Grade 1 (post-baseline) | 1
  Hemoglobin increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  INR increased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 1
  INR increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 1
  Leukocytosis: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Lymphocyte count decreased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Lymphocyte count increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Neutrophil count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Neutrophil count decreased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Platelet count decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Platelet count decreased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  White blood cell decreased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  White blood cell decreased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1

25. Secondary Outcome: Number of Participants With Shift From Baseline for Biochemistry Laboratory Test Abnormalities Based on NCI-CTCAE v4.03: Phase 2
Description: Biochemistry laboratory test included: alanine aminotransferase increased, alkaline phosphatase increased, aspartate aminotransferase increased, blood bilirubin increased, CK increased, creatinine increased, hypercalcemia, hyperglycemia, hyperkalemia, hypermagnesemia, hypernatremia, hypoalbuminemia, hypocalcemia, hypoglycemia, hypokalemia, hypomagnesemia, hyponatremia, hypophosphatemia, lipase increased, and serum amylase increased. Laboratory results were categorically summarized according to the NCI-CTCAE criteria v4.03. Grade 1= mild; Grade 2= moderate; Grade 3= severe and Grade 4= life-threatening or disabling. Grade 0 was assigned for all non-missing values not graded as 1 or higher per CTCAE criteria. Number of participants with shift from baseline for biochemistry laboratory test were assessed. Only those laboratory test parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: as for outcome 24
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 1
  Alanine aminotransferase increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline) | 1
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 4 (post-baseline): number analyzed (Participants) | 2
  Alanine aminotransferase increased: Grade 1 (baseline) to Grade 4 (post-baseline) | 1
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 1
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Alkaline phosphatase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Alkaline phosphatase increased: Grade 2 (baseline) to Grade 2 (post-baseline): number analyzed (Participants) | 1
  Alkaline phosphatase increased: Grade 2 (baseline) to Grade 2 (post-baseline) | 1
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline): number analyzed (Participants) | 2
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 3 (post-baseline): number analyzed (Participants) | 2
  Aspartate aminotransferase increased: Grade 0 (baseline) to Grade 3 (post-baseline) | 1
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 1
  Aspartate aminotransferase increased: Grade 1 (baseline) to Grade 0 (post-baseline) | 1
  Blood bilirubin increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  CK increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  CK increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 1
  Creatinine increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Creatinine increased: Grade 0 (baseline) to Grade 2 (post-baseline) | 2
  Hypercalcemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hyperglycemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hyperkalemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hypermagnesemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hypernatremia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hypoalbuminemia: Grade 0 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 2
  Hypoalbuminemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Hypoalbuminemia: Grade 1 (baseline) to Grade 0 (post-baseline): number analyzed (Participants) | 1
  Hypoalbuminemia: Grade 1 (baseline) to Grade 0 (post-baseline) | 1
  Hypocalcemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 1
  Hypocalcemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 2
  Hypoglycemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hypokalemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Hypokalemia: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Hypomagnesemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hyponatremia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Hypophosphatemia: Grade 0 (baseline) to Grade 0 (post-baseline) | 3
  Lipase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Lipase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1
  Serum amylase increased: Grade 0 (baseline) to Grade 0 (post-baseline) | 2
  Serum amylase increased: Grade 0 (baseline) to Grade 1 (post-baseline) | 1

26. Secondary Outcome: Number of Participants With Clinically Significant Change in Notable Abnormal Vital Signs: Phase 2
Description: In this outcome measure, number of participants with notable abnormal vital signs included: systolic and diastolic BP in mmHg based on following criteria: 1) High Systolic BP: >=160 mmHg and an increase >=20 mmHg from baseline; 2) High Diastolic BP: >=100 mmHg and an increase >=15 mmHg from baseline; 3) Low Systolic BP: <=90 mmHg with decrease from baseline of >=20 mmHg; 4) Low Diastolic BP: <=50 mmHg with decrease from baseline of >=15 mmHg; pulse rate in bpm based on following criteria: 1) High pulse rate >=120 bpm with increase from baseline of >=15 bpm; 2) Low pulse rate <=50 bpm with decrease from baseline of >=15 bpm; weight in kg based on following criteria: 1) Weight: Increase from baseline of >=10%, 2) Weight: >=20 % decrease from baseline; temperature in degree C based on following criteria: 1) High body temperature >=37.5 degree C, 2) Low body temperature <=36 degree C. Only those vital signs parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants
  Increased body weight | 1
  Low body temperature | 2

27. Secondary Outcome: Number of Participants With Notable Abnormal Electrocardiogram (ECG) Values: Phase 2
Description: In this outcome measure, number of participants with notable abnormal ECG values included: QTcF values in msec based on following criteria: 1) increase from baseline >30 msec; 2) increase from baseline >60 msec; 3) new >450 msec; 4) new >480 msec; and 5) new >500 msec; heart rate values in bpm based on following criteria: 1) Increase from baseline >25% and to a value >100; 2) Decrease from baseline >25% and to a value <50. Only those vital ECG parameters in which at least 1 participant had data were reported.
Time Frame: Baseline (Day 1) up to 30 days after last dose of study drug in Phase 2, maximum duration up to 8.3 months
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
Number analyzed (Participants) | 3
Participants | 1

28. Secondary Outcome: Plasma Concentrations of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, plasma concentrations (in nanogram per milliliter [ng/mL]) of encorafenib and its metabolite LHY746 at Cycle 1 Day 1 (C1D1), Cycle 1 Day 15 (C1D15), Cycle 2 Day 1 (C2D1), and Cycle 3 Day 1 (C3D1) at different time points were reported.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose; Pre-dose on Cycle 2 Day 1, Cycle 3 Day 1
Population: The pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of any study drug and had at least 1 PK blood collection after the first dose of study drug with associated bioanalytical results. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at specified time points. This outcome measure was planned to be analyzed in SLI phase only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng/mL
  Encorafenib C1D1: 0.5 hrs post dose | 65.5 (328.8)
  Encorafenib C1D1: 1.5 hrs post dose | 1830 (325.5)
  Encorafenib C1D1: 3 hrs post dose | 2120 (36.3)
  Encorafenib C1D1: 6 hrs post dose: number analyzed (Participants) | 7
  Encorafenib C1D1: 6 hrs post dose | 1170 (67.7)
  Encorafenib C1D15: pre-dose: number analyzed (Participants) | 6
  Encorafenib C1D15: pre-dose | 92.3 (87.9)
  Encorafenib C1D15: 0.5 hrs post dose: number analyzed (Participants) | 6
  Encorafenib C1D15: 0.5 hrs post dose | 182 (243.5)
  Encorafenib C1D15: 1.5 hrs post dose: number analyzed (Participants) | 6
  Encorafenib C1D15: 1.5 hrs post dose | 745 (132.7)
  Encorafenib C1D15: 3 hrs post dose: number analyzed (Participants) | 6
  Encorafenib C1D15: 3 hrs post dose | 953 (50.0)
  Encorafenib C1D15: 6 hrs post dose: number analyzed (Participants) | 6
  Encorafenib C1D15: 6 hrs post dose | 332 (61.0)
  Encorafenib C2D1: pre-dose: number analyzed (Participants) | 4
  Encorafenib C2D1: pre-dose | 59.7 (65.7)
  Encorafenib C3D1: pre-dose: number analyzed (Participants) | 5
  Encorafenib C3D1: pre-dose | 50.1 (47.8)
  LHY746 C1D1: 0.5 hrs post dose | 6.46 (114.1)
  LHY746 C1D1: 1.5 hrs post dose | 123 (345.5)
  LHY746 C1D1: 3 hrs post dose: number analyzed (Participants) | 6
  LHY746 C1D1: 3 hrs post dose | 296 (46.7)
  LHY746 C1D1: 6 hrs post dose: number analyzed (Participants) | 7
  LHY746 C1D1: 6 hrs post dose | 277 (62.7)
  LHY746 C1D15: pre-dose: number analyzed (Participants) | 6
  LHY746 C1D15: pre-dose | 892 (101.1)
  LHY746 C1D15: 0.5 hrs post dose: number analyzed (Participants) | 6
  LHY746 C1D15: 0.5 hrs post dose | 941 (88.2)
  LHY746 C1D15: 1.5 hrs post dose: number analyzed (Participants) | 6
  LHY746 C1D15: 1.5 hrs post dose | 1040 (93.4)
  LHY746 C1D15: 3 hrs post dose | 1690 (64.3)
  LHY746 C1D15: 6 hrs post dose: number analyzed (Participants) | 6
  LHY746 C1D15: 6 hrs post dose | 1520 (59.0)
  LHY746 C2D1: pre-dose: number analyzed (Participants) | 4
  LHY746 C2D1: pre-dose | 655 (91.3)
  LHY746 C3D1: pre-dose: number analyzed (Participants) | 5
  LHY746 C3D1: pre-dose | 256 (2956.0)

29. Secondary Outcome: Plasma Concentrations of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, plasma concentrations of binimetinib and its metabolite AR00426032 at C1D1, C1D15, C2D1, and C3D1 at different time points were reported.
Time Frame: as for outcome 28
Population: The PK set included all participants who received at least 1 dose of any study drug and had at least 1 PK blood collection after the first dose of study drug with associated bioanalytical results. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable at specified time points. This outcome measure was planned to be analyzed in SLI phase only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng/mL
  Binimetinib C1D1: 0.5 hrs post dose | 86.6 (567.4)
  Binimetinib C1D1: 1.5 hrs post dose | 297 (341.9)
  Binimetinib C1D1: 3 hrs post dose | 233 (83.2)
  Binimetinib C1D1: 6 hrs post dose: number analyzed (Participants) | 7
  Binimetinib C1D1: 6 hrs post dose | 151 (91.6)
  Binimetinib C1D15: pre-dose: number analyzed (Participants) | 6
  Binimetinib C1D15: pre-dose | 47.7 (71.8)
  Binimetinib C1D15: 0.5 hrs post dose: number analyzed (Participants) | 6
  Binimetinib C1D15: 0.5 hrs post dose | 151 (67.8)
  Binimetinib C1D15: 1.5 hrs post dose: number analyzed (Participants) | 6
  Binimetinib C1D15: 1.5 hrs post dose | 232 (121.1)
  Binimetinib C1D15: 3 hrs post dose: number analyzed (Participants) | 6
  Binimetinib C1D15: 3 hrs post dose | 215 (55.2)
  Binimetinib C1D15: 6 hrs post dose: number analyzed (Participants) | 6
  Binimetinib C1D15: 6 hrs post dose | 79.9 (56.6)
  Binimetinib C2D1: pre-dose: number analyzed (Participants) | 4
  Binimetinib C2D1: pre-dose | 42.0 (47.8)
  Binimetinib C3D1: pre-dose: number analyzed (Participants) | 5
  Binimetinib C3D1: pre-dose | 30.0 (65.3)
  AR00426032 C1D1: 0.5 hrs post dose | 8.10 (132.4)
  AR00426032 C1D1: 1.5 hrs post dose | 30.3 (345.7)
  AR00426032 C1D1: 3 hrs post dose | 31.7 (60.1)
  AR00426032 C1D1: 6 hrs post dose: number analyzed (Participants) | 7
  AR00426032 C1D1: 6 hrs post dose | 21.9 (36.6)
  AR00426032 C1D15: pre-dose: number analyzed (Participants) | 6
  AR00426032 C1D15: pre-dose | 3.13 (53.0)
  AR00426032 C1D15: 0.5 hrs post dose: number analyzed (Participants) | 6
  AR00426032 C1D15: 0.5 hrs post dose | 5.89 (136.9)
  AR00426032 C1D15: 1.5 hrs post dose: number analyzed (Participants) | 6
  AR00426032 C1D15: 1.5 hrs post dose | 10.6 (56.8)
  AR00426032 C1D15: 3 hrs post dose: number analyzed (Participants) | 6
  AR00426032 C1D15: 3 hrs post dose | 12.5 (58.0)
  AR00426032 C1D15: 6 hrs post dose: number analyzed (Participants) | 6
  AR00426032 C1D15: 6 hrs post dose | 4.71 (62.8)
  AR00426032 C2D1: pre-dose: number analyzed (Participants) | 4
  AR00426032 C2D1: pre-dose | 2.97 (29.6)
  AR00426032 C3D1: pre-dose: number analyzed (Participants) | 5
  AR00426032 C3D1: pre-dose | 1.57 (42.2)

30. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 6 Hours (AUC 0-6) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, area under the plasma concentration-time curve from zero to 6 hours (AUC 0-6) after administration of encorafenib and its metabolite LHY746 in nanogram*hour per milliliter (ng*hr/mL) at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 7
ng*hr/mL
  Encorafenib: C1D1 | 9530 (50.6)
  Encorafenib: C1D15: number analyzed (Participants) | 6
  Encorafenib: C1D15 | 3930 (52.8)
  LHY746: C1D1 | 1230 (60.1)
  LHY746: C1D15: number analyzed (Participants) | 6
  LHY746: C1D15 | 8160 (67.7)

31. Secondary Outcome: AUC0-6 of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, area under the plasma concentration-time curve from zero to 6 hours (AUC 0-6) after administration of binimetinib and its metabolite AR00426032 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 7
ng*hr/mL
  Binimetinib: C1D1 | 1410 (85.5)
  Binimetinib: C1D15: number analyzed (Participants) | 6
  Binimetinib: C1D15 | 1050 (39.7)
  AR00426032: C1D1 | 159 (65.9)
  AR00426032: C1D15: number analyzed (Participants) | 6
  AR00426032: C1D15 | 53.9 (48.6)

32. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Last Time Point (AUClast) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, area under the plasma concentration-time curve from zero to the last measurable time point (AUClast) after administration of encorafenib and its metabolite LHY746 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng*hr/mL
  Encorafenib: C1D1 | 9190 (47.8)
  Encorafenib: C1D15: number analyzed (Participants) | 6
  Encorafenib: C1D15 | 7490 (52.8)
  LHY746: C1D1 | 1180 (56.9)
  LHY746: C1D15: number analyzed (Participants) | 6
  LHY746: C1D15 | 29600 (73.0)

33. Secondary Outcome: AUClast of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, area under the plasma concentration-time curve from zero to the last measurable time point (AUClast) after administration of binimetinib and its metabolite AR00426032 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng*hr/mL
  Binimetinib: C1D1 | 1350 (79.1)
  Binimetinib: C1D15: number analyzed (Participants) | 6
  Binimetinib: C1D15 | 1440 (43.9)
  AR00426032: C1D1 | 156 (60.6)
  AR00426032: C1D15: number analyzed (Participants) | 6
  AR00426032: C1D15 | 77.9 (49.7)

34. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Tau (AUCtau) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, area under the plasma concentration-time curve from time zero to the last measurable time point Tau (AUCtau) of encorafenib and its metabolite LHY746 over a dosing interval (6 hours as appropriate) of C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: The PK set included all participants who received at least 1 dose of any study drug and had at least 1 PK blood collection after the first dose of study drug with associated bioanalytical results. Here 'Overall Number of Participants Analyzed' signifies number of participants evaluable for this outcome measure. This outcome measure was planned to be analyzed in SLI phase only.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng*hr/mL
  Encorafenib | 7490 (52.8)
  LHY746 | 29600 (73.0)

35. Secondary Outcome: AUCtau of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: as for outcome 34
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng*hr/mL
  Binimetinib | 1440 (43.9)
  AR00426032 | 77.9 (49.7)

36. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) After Drug Administration of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, maximum observed plasma concentration (Cmax) after administration of encorafenib and its metabolite LHY746 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng/mL
  Encorafenib: C1D1 | 3210 (47.7)
  Encorafenib: C1D15: number analyzed (Participants) | 6
  Encorafenib: C1D15 | 1370 (79.3)
  LHY746: C1D1 | 340 (47.2)
  LHY746: C1D15: number analyzed (Participants) | 6
  LHY746: C1D15 | 1720 (65.3)

37. Secondary Outcome: Cmax of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, maximum observed plasma concentration (Cmax) after administration of binimetinib and its metabolite AR00426032 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ng/mL
  Binimetinib: C1D1 | 506 (85.5)
  Binimetinib: C1D15: number analyzed (Participants) | 6
  Binimetinib: C1D15 | 359 (40.5)
  AR00426032: C1D1 | 53.9 (77.8)
  AR00426032: C1D15: number analyzed (Participants) | 6
  AR00426032: C1D15 | 16.9 (54.0)

38. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) at the End of a Dosing Interval at Steady State of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, minimum observed plasma concentration (Cmin) after administration of encorafenib and its metabolite LHY746 at C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng/mL
  Encorafenib | 91.1 (88.3)
  LHY746 | 829 (99.3)

39. Secondary Outcome: Cmin of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, minimum observed plasma concentration (Cmin) after administration of binimetinib and its metabolite AR00426032 at C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng/mL
  Binimetinib | 47.7 (71.8)
  AR00426032 | 3.04 (47.8)

40. Secondary Outcome: Ctrough of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, measured concentration at the end of a dosing interval (Ctrough) of encorafenib and its metabolite LHY746 at C1D15 were assessed.
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng/mL
  Encorafenib | 332 (61.0)
  LHY746 | 1520 (59.0)

41. Secondary Outcome: Ctrough of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, measured concentration at the end of a dosing interval (Ctrough) of binimetinib and its metabolite AR00426032 at C1D15 were assessed.
Time Frame: as for outcome 28
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ng/mL
  Binimetinib | 79.9 (56.6)
  AR00426032 | 4.71 (62.8)

42. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, time to reach maximum concentration (Tmax) of encorafenib and its metabolite LHY746 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hours
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
hours
  Encorafenib: C1D1 | 1.53 [1.47 to 3.00]
  Encorafenib: C1D15: number analyzed (Participants) | 6
  Encorafenib: C1D15 | 1.55 [0.43 to 3.00]
  LHY746: C1D1 | 4.33 [1.47 to 6.00]
  LHY746: C1D15: number analyzed (Participants) | 6
  LHY746: C1D15 | 3.00 [2.92 to 5.73]

43. Secondary Outcome: Tmax of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, time to reach maximum concentration (Tmax) of binimetinib and its metabolite AR00426032 at C1D1, and C1D15 were assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hrs (+/- 20 minutes [min]) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs (+/- 20 min) post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hours
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
hours
  Binimetinib: C1D1 | 1.50 [1.45 to 6.08]
  Binimetinib: C1D15: number analyzed (Participants) | 6
  Binimetinib: C1D15 | 1.55 [0.43 to 2.98]
  AR00426032: C1D1 | 1.53 [1.47 to 6.08]
  AR00426032: C1D15: number analyzed (Participants) | 6
  AR00426032: C1D15 | 1.58 [0.43 to 3.07]

44. Secondary Outcome: Time of Last PK Sample (Tlast) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, time of last PK sample (Tlast) of encorafenib and its metabolite LHY746 at C1D1, and C1D15 were assessed. As outlined in the prespecified Statistical Analysis Plan for the study, since encorafenib was administered in continuous cycles, the pre-dose sample on Cycle 2 Day 1 was assumed to be at steady state and was interpolated as the concentration on 24 hours for encorafenib and LHY746 on Cycle 1 Day 15 during the analysis. In doing so, the reported Tlast values from the noncompartmental analysis (NCA) are 24 hours for encorafenib and LHY746.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6, 24 hrs post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hours
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
hours
  Encorafenib: C1D1 | 5.78 [3.00 to 6.08]
  Encorafenib: C1D15: number analyzed (Participants) | 6
  Encorafenib: C1D15 | 24.00 [24.00 to 24.00]
  LHY746: C1D1 | 5.78 [3.00 to 6.08]
  LHY746: C1D15: number analyzed (Participants) | 6
  LHY746: C1D15 | 24.00 [24.00 to 24.00]

45. Secondary Outcome: Tlast of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, time of last PK sample (Tlast) of binimetinib and its metabolite AR00426032 at C1D1, and C1D15 were assessed. As outlined in the prespecified Statistical Analysis Plan for the study, since binimetinib was administered in continuous cycles, the pre-dose sample on Cycle 2 Day 1 was assumed to be at steady state and was interpolated as the concentration for 12 hours for binimetinib and AR00426032 on Cycle 1 Day 15 for the noncompartmental analysis. In doing so, the reported Tlast values from the noncompartmental analysis (NCA) are 12 hours for binimetinib and AR00426032.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6, 12 hrs post-dose
Population: as for outcome 29
Measure: Median (Full Range); unit: hours
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
hours
  Binimetinib: C1D1 | 5.78 [3.00 to 6.08]
  Binimetinib: C1D15: number analyzed (Participants) | 6
  Binimetinib: C1D15 | 12.00 [12.00 to 12.00]
  AR00426032: C1D1 | 5.78 [3.00 to 6.08]
  AR00426032: C1D15: number analyzed (Participants) | 6
  AR00426032: C1D15 | 12.00 [12.00 to 12.00]

46. Secondary Outcome: Accumulation Ratio Between AUClast,ss and AUClast (RAUC) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, accumulation ratio of encorafenib and its metabolite LHY746 calculated as: C1D15 AUC0-6 divided by C1D1 AUC0-6 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ratio
  Encorafenib | 0.468 (46.0)
  LHY746 | 7.25 (46.7)

47. Secondary Outcome: RAUC of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, accumulation ratio of binimetinib and its metabolite AR00426032 calculated as: C1D15 AUC0-6 divided by C1D1 AUC0-6 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ratio
  Binimetinib | 0.877 (60.4)
  AR00426032 | 0.359 (93.0)

48. Secondary Outcome: Accumulation Ratio Between Cmax,ss and Cmax (RCmax) of Encorafenib and Its Metabolite LHY746: SLI Phase
Description: In this outcome measure, accumulation ratio of encorafenib and its metabolite LHY746 calculated as: C1D15 Cmax divided by C1D1 Cmax was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ratio
  Encorafenib | 0.490 (71.8)
  LHY746 | 5.78 (41.7)

49. Secondary Outcome: Rcmax of Binimetinib and Its Metabolite AR00426032: SLI Phase
Description: In this outcome measure, accumulation ratio of binimetinib and its metabolite AR00426032 calculated as: C1D15 Cmax divided by C1D1 Cmax was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 34
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 6
ratio
  Binimetinib | 0.818 (95.9)
  AR00426032 | 0.347 (130.9)

50. Secondary Outcome: Ratio of AUClast Values of the Metabolite Compared to Parent (MRAUClast) of LHY746: SLI Phase
Description: In this outcome measure, ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, for LHY746/encorafenib at C1D1, and C1D15 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 7
ratio
  C1D1 | 0.164 (21.7)
  C1D15: number analyzed (Participants) | 6
  C1D15 | 2.64 (36.0)

51. Secondary Outcome: MRAUClast of AR00426032: SLI Phase
Description: In this outcome measure, ratio of AUClast values of the metabolite compared to parent, corrected for molecular weight, for AR00426032/binimetinib at C1D1, and C1D15 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 7
ratio
  C1D1 | 0.109 (54.1)
  C1D15: number analyzed (Participants) | 6
  C1D15 | 0.0494 (63.9)

52. Secondary Outcome: Ratio of Cmax Values of the Metabolite Compared to Parent (MRCmax) of LHY746: SLI Phase
Description: In this outcome measure, ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, for LHY746/encorafenib at C1D1, and C1D15 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ratio
  C1D1 | 0.135 (16.7)
  C1D15: number analyzed (Participants) | 6
  C1D15 | 1.59 (47.8)

53. Secondary Outcome: MRCmax of AR00426032: SLI Phase
Description: In this outcome measure, ratio of Cmax values of the metabolite compared to parent, corrected for molecular weight, for AR00426032/ binimetinib at C1D1, and C1D15 was assessed.
Time Frame: Cycle 1 Day 1: 0.5, 1.5, 3, 6 hours (hrs) post-dose; Cycle 1 Day 15: Pre-dose, 0.5, 1.5, 3, 6 hrs post-dose
Population: as for outcome 29
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID
Number analyzed (Participants) | 8
ratio
  C1D1 | 0.103 (49.3)
  C1D15: number analyzed (Participants) | 6
  C1D15 | 0.0453 (53.8)

ADVERSE EVENTS:
Time Frame: Day 1 of dosing up to 30 days after last dose of study drug in Safety Lead-in Phase (maximum up to 10.4 months) and Phase 2 (maximum up to 8.3 months)
Description: Same event may appear as both an AE and SAE. However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID
All-Cause Mortality (participants affected / at risk) | 7/10 | 3/3
Serious Adverse Events (participants affected / at risk) | 4/10 | 1/3
Other Adverse Events (participants affected / at risk) | 10/10 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID (N=10) | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID (N=3)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Air embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Lead-in Phase: Encorafenib 300 mg BID + Binimetinib 45 mg BID (N=10) | Phase 2, Standard Dose Arm: Encorafenib 450 mg QD + Binimetinib 45 mg BID (N=3)
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Macular oedema (Eye disorders) | 0 | 1
Retinopathy (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Facial pain (General disorders) | 1 | 0
Fatigue (General disorders) | 6 | 1
Influenza like illness (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 0
Bronchitis (Infections and infestations) | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 5 | 2
Aspartate aminotransferase increased (Investigations) | 3 | 2
Blood creatine phosphokinase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 2 | 0
Lipase increased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 2 | 0
Transaminases increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Disturbance in attention (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Facial paresis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 0
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 3 | 0
Stress (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 1 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 0
Melanocytic hyperplasia (Skin and subcutaneous tissue disorders) | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
Data for pharmacokinetic outcome measure for "Phase 2" was not collected and analyzed as sampling was insufficient to support noncompartmental analysis in participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/69/NCT03911869/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03911869/SAP_001.pdf